CLINICAL TRIAL: NCT05500794
Title: Evaluation of the Therapeutic Efficacy of a Mindfulness-Based Stress Reduction (MBSR) Program as an Adjuvant Therapy in Patients With Moderate Pruritic Inflammatory Dermatosis (Psoriasis or Atopic Dermatitis)
Brief Title: Meditation in Inflammatory Dermatosis
Acronym: MediDermIn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP211191
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis; Psoriasis; Pruritus
Keywords: Mindfulness; Based Stress Reduction; Psoriasis; Atopic Dermatitis; Pruritus; Inflammatory Cytokines
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis; Pruritus | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR (Mindfulness-Based Stress Reduction) group (Experimental): MBSR (Mindfulness-Based Stress reduction) program : 1 weekly session of 2 hours and a half for 8 weeks, (first and last session: 3 hours) and an optional day of intensive practice of 6 hours, supervised by an MBSR instructor.
  Interventions: Other: MBSR (Mindfulness-Based Stress Reduction)
- Standard group (No Intervention): No intervention in this group which will be followed according to the standard care

INTERVENTIONS:
Other: MBSR (Mindfulness-Based Stress Reduction) — MBSR (Mindfulness-Based Stress reduction) program : 1 weekly session of 2 hours and a half for 8 weeks, (first and last session: 3 hours) and an optional day of intensive practice of 6 hours, supervised by an MBSR instructor.
  In each weekly session, the instructor creates a supportive environment in which:
  * Guided meditation practices;
  * Mindfulness stretching and yoga;
  * Reflection and group discussion periods aimed at promoting mindfulness in daily life;
  * Practice instructions and opportunity to ask questions;
  * Instructions for home practice. Audio recordings and a manual are provided to support personal practice.
  Audio recordings and a manual are provided to support personal practice
  Arms: MBSR (Mindfulness-Based Stress Reduction) group

SUMMARY:
Psoriasis and atopic dermatitis are multifactorial inflammatory dermatoses, with a very high prevalence, reaching more than 120 million patients in the world. Although the physiopathological mechanisms are not yet clearly defined, these inflammatory dermatoses involve an interaction between the immune system and the epidermal cells, severe skin inflammation and often very intense pruritus. The objectives of an effective management should be to treat lesions in order to reduce them, but also to reduce itching and allow the patients to accept and cope with their pathology, without neglecting an improvement in the "Dermatology Life Quality Index" (DLQI) and in the psychological state, sometimes depressive, of the patient. Itching is defined as "a feeling that needs to be scratched urgently" and can cause significant distress along with pain. It severely impacts the quality of life and the quality of sleep. Chronic itching is associated with increased stress, anxiety, and other mood disorders. In turn, stress and anxiety exacerbate the itching, leading to a vicious cycle of pruritus - scratching that affects patient behavior (excessive scratching) and worsens disease prognosis and quality of life. Much research over the past few decades has demonstrated the effect of mindfulness meditation on emotional and cognitive responsiveness, cognitive flexibility, rumination, self-compassion and mindfulness, but also on acute pain, anxiety, stress, depression, cardiovascular disease, eating disorders, cancer and cognitive loss with age. Several studies have shown the impact of mindfulness on brain function and immunity, with evidence for the association between mindfulness and changes in the levels of markers characteristic of immune system activity and inflammation, known to be increased in psoriasis or atopic dermatitis. The objective is to evaluate the effect of mental training in the regulation of stress and emotions through mindfulness meditation in patients with moderate, itchy atopic dermatitis or psoriasis, not treated with systemic agents (e.g.: biotherapies). This project is based on the premise that mental training in the regulation of stress and emotions through meditation would reduce the effects of the infernal itch-scratch cycle, alleviating pruritus, thus improving the well-being and mental health of patients while reducing their inflammatory skin lesions and limiting the appearance of new lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years old or older
* With health insurance coverage
* Significant pruritus defined by a Visual Analogical Scale (VAS) pruritus ≥ 4
* Patient with plaque psoriasis

  * Without joint involvement
  * Mild to moderate severity (PASI>10)
  * DLQI > 10

OR Patient with atopic dermatitis:

* Mild to moderate severity (SCORAD>10)
* DLQI > 10
* Diagnosis according to Hanifin and Raijka criteria

  * Patient in a stable psychological state
  * French langage spoken

Exclusion Criteria :

* Current systemic treatment or treatment discontinued within the last month
* Psychiatric illnesses diagnosed according to the DSM-5 or ICD-10 international criteria of psychotic disorder, severe anxiety disorder, depressive disorder with a current depressive episode of severe intensity, bipolar disorder with a current depressive or manic episode
* Taking psychotropic or neuroleptic treatments
* Participation in another interventional research study or being in the exclusion period at the end of a previous study, if applicable
* Patient under AME

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Pruritus assessed by Visual Analogue Scale (VAS) | at 8 weeks
  VAS Pruritus scale is a scale going from 0 to 10. 0 corresponds to no pruritus et 10 to the maximum of prurit.

SECONDARY OUTCOMES:
Pruritus assessed by Visual Analogue Scale (VAS) | at 16 weeks
  VAS Pruritus scale is a scale going from 0 to 10. 0 corresponds to no pruritus et 10 to the maximum of prurit.
Pruritus assessed by 5-D Itch Scale 5-D (5-D IQ) | at 8 weeks
  The 5-D itch scale is a multidimensional questionnaire. The scores of each of the domains are achieved separately and then summed together : total 5-D score can potentially range between 5 (no pruritus) and 25 (most severe pruritus).
Pruritus assessed by 5-D Itch Scale 5-D (5-D IQ) | at 16 weeks as compared to 8 weeks
  The 5-D itch scale is a multidimensional questionnaire. The scores of each of the domains are achieved separately and then summed together : total 5-D score can potentially range between 5 (no pruritus) and 25 (most severe pruritus).
Number of dermatocorticoides tubes | at 8 weeks
Number of dermatocorticoides tubes | at 16 weeks as compared to 8 weeks
Number of scratches per day (including nights) | at 8 weeks
Number of scratches per day (including nights) | at 16 weeks as compared to 8 weeks
Psorasis Area and severity index (PASI Index) for psoriasis group | at 8 weeks
  This score takes into account the affected skin surface, the degree of redness, the thickening of the skin and the scaling. Its ranges from 0 to 72.The higher the number, the more severe the psoriasis.
Psorasis Area and severity index (PASI Index) for psoriasis group | at 16 weeks as compared to 8 weeks
  This score takes into account the affected skin surface, the degree of redness, the thickening of the skin and the scaling. Its ranges from 0 to 72.The higher the number, the more severe the psoriasis.
SCORAD Index for atopic dermatitis | at 8 weeks
  The maximal score of the SCORAD Index is 103.
SCORAD Index for atopic dermatitis | at 16 weeks as compared to 8 weeks
  The maximal score of the SCORAD Index is 103.
Stress evaluation assessed by Perceived Stress Scale | at 8 weeks
  It is a 10 questions scale with 5 items per question. Its goes from 10 to 50.
Stress evaluation assessed by Perceived Stress Scale | at 16 weeks as compared to 8 weeks
  It is a 10 questions scale with 5 items per question. Its goes from 10 to 50.
Quantification of inflammatory stress markers in saliva | at 8 weeks
  Saliva stress markers will be alpha-amylase, cortisol, IL-6, IL-31 and TNF-alpha
Quantification of inflammatory stress markers in saliva | at 16 weeks as compared to 8 weeks
  Saliva stress markers will be alpha-amylase, cortisol, IL-6, IL-31 and TNF-alpha
Quantification of inflammatory stress markers in serum | at 8 weeks
  Serum stress markers will be CRP, cortisol, IL-6, IL-3, TNF-alpha and Adreno CorticoTropic Hormone
Quantification of inflammatory stress markers in serum | at 16 weeks as compared to 8 weeks
  Serum stress markers will be CRP, cortisol, IL-6, IL-31,TNF-alpha and Adreno CorticoTropic Hormone

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint-Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided